CLINICAL TRIAL: NCT05386537
Title: Combining Wearable Robotic Orthosis With Visual and Haptic Feedback to Enhance the Recovery of Upper Extremity Motor Function and ADL in Persons With Acute SCI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D-1113-20
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- MyoPro-VR/HM group (Experimental): Receive 18 sessions (in 6 weeks) of wrist/hand/UE rehabilitation using the MyoPro wearable robotic orthosis combined with VR-video games and Haptics.
  Interventions: Combination Product: MyoMo orthosis and VR games; Device: MyoPro robot only; Other: Games only
- MyoPro group (Active Comparator): Receive 18 sessions (in 6 weeks) of wrist/hand/UE rehabilitation using the MyoPro wearable robotic orthosis only.
  Interventions: Device: MyoPro robot only
- VR/HM group (Active Comparator): Receive 18 sessions (in 6 weeks) of wrist/hand/UE rehabilitation using VR-video games only.
  Interventions: Other: Games only
- control (Other): Receive 18 sessions (in 6 weeks) of conventional UE therapy at a rehabilitation facility.
  Interventions: Other: Control

INTERVENTIONS:
Combination Product: MyoMo orthosis and VR games — Combining Wearable Robotic Orthosis with Visual and Haptic Feedback to Enhance the Recovery of Upper Extremity Motor Function and ADL in Persons with Acute SCI
  Other Names: Control
  Arms: MyoPro-VR/HM group
Device: MyoPro robot only — Using the MyoPro wearable robotic orthosis only
  Arms: MyoPro group; MyoPro-VR/HM group
Other: Games only — Using VR-video games only
  Arms: MyoPro-VR/HM group; VR/HM group
Other: Control — conventional UE therapy at a rehabilitation facility
  Arms: control

SUMMARY:
This randomized clinical trial (RCT) is evaluating the usefulness of combining MyoMo robotic orthosis with visual and haptic feedback in ameliorating wrist/hand/UE movement capability, and increasing ADL and quality of life in people with acute SCI.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-80
* Be able to activate the muscles of my upper arm and forearm with enough strength as determined by the therapist.
* Be diagnosed with a spinal cord injury (iSCI (ASIA Impairment Scale (AIS) C and D) and be less than 3 months post initial injury at the start of the study
* Be medically stable
* Be able to follow study directions and communicate in English as determined by the study staff
* Continue to take all prescribed medication (example: baclofen: oral or via pump) without any major dosing changes
* Be able to tolerate functional tasks for 60min with intermittent rests without excessive fatigue
* Have full passive range of motion at my elbow, as determined by study staff

Exclusion Criteria:

* Be younger than 18 years old or older than 80
* Have excessive pain in my arm or hand that would limit my participation in rehabilitation
* Have excessive spasticity in my elbow or wrist joints as determined by study staff
* Be participating in any experimental rehabilitation or drug studies
* Have a history of neurologic disorder other than spinal cord injury
* Have other conditions that would prevent safe and/or effective participation using the study device. Examples of these conditions include: severe sensory deficits, skin conditions, joint contractures, etc.
* Have difficulty following multiple step directions
* Have severe psychiatric problems or difficulty thinking clearly that would prevent me from participating in this study
* Have skin issues that would prevent wearing the Myo-Pro device
* Have had history of recurrent epilepsy, seizure or convulsion
* Have a past or current history of treated ringing in the ears known as tinnitus or severe hearing problems.
* Be taking any drugs that would increase my risk of having a seizure while undergoing brain stimulation. Study staff and physician will review my medications to see if I am taking any of these drugs. If I am taking one of these drugs, I will not be enrolled in this study.
* Because of potential risk to the fetus, women of child-bearing potential will be required to have a pregnancy test before they can enroll in this study. If I am female, and have a positive pregnancy test, I will not be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Range of motion of hands and arms | Approximately 10 weeks
  Movement of upper extremity is measured using small sensors that are able to record joints' angles. These sensors are placed on participant's skin via double sticky tape.
  Participants will be asked to move their hand and forearm while the elbow, wrist and hand joint angles are measured.
Muscle strength measurement | Approximately 10 weeks
  during movements of upper extremities muscle strength is measured using small and light weight surface electromyography sensors which are placed on the participant's skin via double stick tape.
  Participants will be asked to move their hand and forearm while the muscle strength is measured.
GRASSP | Approximately 10 weeks
  Assessment of the Hand in Tetraplegia Using the Graded Redefined Assessment of Strength Sensibility and Prehension Upper Extremity Function in Persons with Tetraplegia Relationships Between Strength, Capacity and the Spinal Cord Independence Measure.
  Total score's minimum and maximum values are between 0 to 116 and higher scores indicate better/improved outcomes.

SECONDARY OUTCOMES:
Brain signals measurement | Approximately 10 weeks
  Measurements of brain signals is done using a cap and electrodes that would be placed on the participant's head using surface electrodes.
  Participants will be asked to move their extremities while brain signals are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided